CLINICAL TRIAL: NCT04818125
Title: Circulating Cancer Cells/Macrophage HYbrid Cells in Patients With Breast Cancer.
Acronym: CARMMYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21 SEIN 01
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer cell/macrophage hybrid cells; Hybrid cells
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with breast cancer (Other)
  Interventions: Other: Patients with breast cancer (stage I, II III or IV)

INTERVENTIONS:
Other: Patients with breast cancer (stage I, II III or IV) — Blood samples will be collected at different times:
  * at Baseline for all patients with breast cancer: before initiation of treatment (i.e. before initiation of planned treatment for stage I to III patients and before any new line of treatment for stage IV patients);
  * at the time of disease progression (or at 12 months in absence of progression) for patients with metastatic breast cancer (stage IV)
  For each patient a tumor sample from the initial diagnosis of the disease (i.e. primary tumor +/- biopsy of a metastasis) will be collected (archived tumor block) for the study.

SUMMARY:
Pilot, prospective, monocentric study aimed at evaluating the rate of patients with circulating cancer cell/macrophage hybrid cells in the peripheral blood.

The study will be conducted on a population of patients with breast cancer (regardless of stage of the disease and the immunohistochemical subtype).

For each included patient, blood samples will be taken and tumor specimens will be collected for the study.

At the end of the blood collection, the patient will have completed his participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with breast cancer of any stage (stage I, II, III or IV) and any immunohistochemical subtype (triple-negative, HR+/HER2-negative or HER2-positive).
2. Patient not yet initiated on specific treatment for the stage of breast cancer at inclusion.
3. Available tumor sample (archived tumor block) : initial tumor or metastasis depending on the stage of the disease and availability.
4. Age ≥ 18 years old.
5. Patient affiliated to a Social Health Insurance in France.
6. Patient having signed informed consent prior to inclusion in the study and prior to any specific study procedure.

Exclusion Criteria:

1. Associated pathology(ies) that may prevent the proper conduct of the procedure under consideration.
2. Pregnant or breastfeeding woman.
3. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures of the study protocol.
4. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship protection of justice).
5. Patient who has presented another solid tumor (except breast or cervix carcinoma in situ) within 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Rate of patients with cancer cell / macrophage hybrid cells in peripheral blood defined as the ratio of the number of patients with hybrid cells to the total number of patients. | 20 months after the study start

SECONDARY OUTCOMES:
Quantification of circulating hybrid cells in peripheral blood by automatic measurement (Cell Counter Corning) and expressed in number of cells / millilitre of blood. | 20 months after the study start
Progression-free survival (PFS) defined as the time from the date of inclusion to the date of progression or death from any cause. | 20 months after the study start

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France